CLINICAL TRIAL: NCT06559982
Title: Effects of a Brown Seaweed Extract and Tart Cherry Blend Cardiometabolic Outcomes in Participants With Mild-moderate Hypertension an Ex-vivo Optimized Pilot Feasibility Trial
Brief Title: Effects of a Brown Seaweed Tart Cherry Blend in Mild-moderate Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Seaweed-cherry hypertension
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Identical in taste and colour to the supplement juice, but with no peppermint content.
  Interventions: Other: Placebo
- Brown seaweed and tart cherry blend (Experimental)
  Interventions: Dietary Supplement: Brown seaweed and tart cherry blend

INTERVENTIONS:
Dietary Supplement: Brown seaweed and tart cherry blend — Blend of brown seaweed and tart cherry blend taken twice daily
  Arms: Brown seaweed and tart cherry blend
Other: Placebo — Identical in taste and colour to the supplement, but with no brown seaweed or tart cherry.
  Arms: Placebo

SUMMARY:
The brown seaweed species Ascophyllum nodosum is rich in bioactive polysaccharides, proteins, peptides, lipids, pigments, and polyphenols. Similarly, Montmorency tart cherry (Prunus cerasus L.) is high in anthocyanins and polyphenols. Both substances have antioxidant, anti-inflammatory, and vasodilatory properties that target mechanisms central to hypertension and cardiometabolic diseases.

Dietary interventions to improve cardiovascular health are highly sought after as they possess less risk and financial burden than pharmacological drugs. Previous randomized trial has shown that both brown seaweed and tart cherry supplementation can improving systolic blood pressure and other cardiovascular/ blood lipids. However, to date, no research has explored a seaweed - tart cherry blend using a placebo randomized intervention in patients with hypertension.

The primary purpose of the proposed investigation is to test the ability of a seaweed - tart cherry supplementation blend to improve cardiometabolic parameters in participants with mild-moderate hypertension using a pilot/ feasibility study.

DETAILED DESCRIPTION:
Hypertension is the leading preventable risk factor for cardiovascular disease and mortality, causing over 75,000 annual UK deaths. It affects 31% of males and 26% of females, with about 30% having uncontrolled blood pressure. The UK has 14.4 million hypertensive individuals due to aging, population growth, and lifestyle factors. Hypertension accounts for 12% of GP appointments and £2.1 billion in annual healthcare costs, making it the most expensive disease modality.

Effective management can significantly reduce stroke and heart disease risk. A 2mmHg reduction in systolic blood pressure decreases coronary heart disease mortality by 7% and stroke risk by 10%. A 5mmHg reduction over 10 years could save the NHS nearly £1 billion. This highlights the need for alternative approaches due to pharmaceutical treatments' high cost and side effects.

The brown seaweed species Ascophyllum nodosum is rich in bioactive polysaccharides, proteins, peptides, lipids, pigments, and polyphenols. Similarly, Montmorency tart cherry (Prunus cerasus L.) is high in anthocyanins and polyphenols. Both substances have antioxidant, anti-inflammatory, and vasodilatory properties that target mechanisms central to hypertension and cardiometabolic diseases. Prior to the commencement of this pilot/ feasibility trial, we will evaluate the efficacy of a brown seaweed-tart cherry blend using an ex-vivo model to determine the optimal proportions of each and to understand the molecular effects. The most bioactive blend will be tested in this trial.

The primary purpose of the proposed investigation is to test the ability of a seaweed - tart cherry supplementation blend to improve cardiometabolic parameters in participants with mild-moderate hypertension using a pilot/ feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18-65 years
* Systolic blood pressure 120 to 139 mmHg
* Not taking prescribed medicine for blood pressure management
* Ability to complete written questionnaires independently
* Able to provide informed consent

Exclusion Criteria:

* Diagnosed with diabetes mellitus and/ or coronary heart disease
* Pregnant and lactating women
* Allergy to peppermint
* Habitual consumption of peppermint products
* Regular consumption of antioxidant supplements
* Body mass index larger than 40.0 kg/m2
* Current enrolment in other clinical trials of other external therapies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Baseline
  Systolic blood pressure - measured using a digital blood pressure monitor
Systolic blood pressure | 20 days
  Systolic blood pressure - measured using a digital blood pressure monitor

SECONDARY OUTCOMES:
Diastolic blood pressure | Baseline
  Diastolic blood pressure - measured using a digital blood pressure monitor
Diastolic blood pressure | 20 days
  Diastolic blood pressure - measured using a digital blood pressure monitor
Percent bodyfat and fat mass | Baseline
  Participants percentage composition of fat - measured using bio-electrical impedance
Percent bodyfat and fat mass | 20 days
  Participants percentage composition of fat - measured using bio-electrical impedance
Waist circumference | Baseline
  Waist circumference - measured using anthropocentric tape
Waist circumference | 20 days
  Waist circumference - measured using anthropocentric tape
Waist to hip ratio | Baseline
  Ratio of waist to hip circumference - measured using anthropocentric tape
Waist to hip ratio | 20 days
  Ratio of waist to hip circumference - measured using anthropocentric tape
Blood glucose | Baseline
  Capillary blood glucose - mmol/L
Blood glucose | 20 days
  Capillary blood glucose - mmol/L
Blood triglycerides | Baseline
  Capillary blood triglycerides - mmol/L
Blood triglycerides | 20 days
  Capillary blood triglycerides - mmol/L
Blood cholesterol (Total, HDL & LDL) | Baseline
  Capillary blood cholesterol - mmol/L
Blood cholesterol (Total, HDL & LDL) | 20 days
  Capillary blood cholesterol - mmol/L
Total and HDL cholesterol ratio | Baseline
  Ratio of total cholesterol to HDL cholesterol
Total and HDL cholesterol ratio | 20 days
  Ratio of total cholesterol to HDL cholesterol
LDL and HDL cholesterol ratio | Baseline
  Ratio of LDL to HDL cholesterol
LDL and HDL cholesterol ratio | 20 days
  Ratio of LDL to HDL cholesterol
Triglyceride glucose index | Baseline
  Log transformed measurement of the blood glucose and blood triglyceride measures
Triglyceride glucose index | 20 days
  Log transformed measurement of the blood glucose and blood triglyceride measures
Coop-Wonka chart | Baseline
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Coop-Wonka chart | 20 days
  Psychological wellbeing - The Coop-Wonka chart is a six item questionnaire with a 1-5 scoring system for each thus the chart has a maximum score of 30 which indicates the lowest possible psychological Wellbeing.
Beck Depression Inventory | Baseline
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
Beck Depression Inventory | 20 days
  Psychological wellbeing - the Beck Depression Inventory is a 21 questionnaire with questions that range in scoring from 0-3, thus the maximum score is 63 which is the highest depression score possible.
State Trait Anxiety Inventory | Baseline
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
State Trait Anxiety Inventory | 20 days
  Psychological wellbeing - the state trait anxiety inventory is a 40 item questionnaire with each question having a 1-4 score system, thus the maximum score is 80 which indicates the highest level of anxiety.
Insomnia Severity Index | Baseline
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Insomnia Severity Index | 20 days
  Sleep quality - The Insomnia Severity Index is a brief instrument designed to assess the severity of both nighttime and daytime components of insomnia. The Insomnia Severity Index is a 7-item self-report questionnaire yielding a total score ranging from 0 to 28.
Pittsburgh Sleep Quality Index | Baseline
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Pittsburgh Sleep Quality Index | 20 days
  Sleep quality - The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.
Epworth Sleepiness Scale | Baseline
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.
Epworth Sleepiness Scale | 20 days
  Sleep quality - The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3) with a maximum score of 24.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided